CLINICAL TRIAL: NCT00841802
Title: Glucocorticosteroid Action in Inflammatory Disease
Brief Title: Chronic Rhinosinusitis With or Without Nasal Polyps Steroid Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Realized there was a design flaw.
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert Schleimer, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00010040; 5R37HL068546 (NIH)
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Chronic Sinusitis; Rhinosinusitis; Nasal Polyps
Keywords: Chronic sinusitis; Chronic rhinosinusitis; Nasal polyps
MeSH Terms: conditions — Rhinosinusitis; Nasal Polyps | interventions — Prednisone; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone (Experimental): Steroid medication
  Interventions: Drug: Prednisone
- No Intervention (No Intervention): No Intervention

INTERVENTIONS:
Drug: Prednisone — Prednisone 30mg once daily x 5 days
  Other Names: Glucocorticoid; Deltasone; Liquid Pred; Meticorten; Orasone; Prednicen-M; Prednicot; Sterapred
  Arms: Prednisone

SUMMARY:
This is a study to evaluate the cause of chronic sinus disease. Oral steroids have long been used in the treatment of inflammatory conditions including chronic sinusitis, asthma, and arthritis. However, it is not well known exactly which patients will benefit from steroids when used in the treatment of chronic sinusitis. For some doctors, it is common practice to use these medications prior to planned sinus surgery, to lessen the inflammation and possibly help the healing process. Other doctors feel oral steroids may not be helpful in this way, and there is no conclusive data as to whether this practice has a long term benefit.

DETAILED DESCRIPTION:
The purpose of this research study is to better understand how this potential treatment option, oral steroids, affects biochemical substances that have been associated with the development of chronic sinusitis and polyps. In order to do this, we need to study people with different forms of chronic sinusitis and compare them to individuals without allergies or sinus disease. We will also look at patients with chronic sinusitis who are treated with oral steroids and compare them to chronic sinus patients who have not received oral steroid therapy prior to surgery. This study may help pave the way to new treatments that address specific parts of the chronic sinus inflammatory pathway.

Hypotheses

1. Oral steroid treatment of patients with CRS will lead to a correction in the inflammation that is observed in sinonasal tissues, nasal brushings, and nasal lavage.
2. Steroid induced changes in inflammation will differ in chronic sinus patients with polyps than in those without polyps.
3. Changes in inflammation will correlate with clinical variables.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years to 70 years
* Diagnosis of chronic rhinosinusitis (CRS) with nasal polyps (NP) and will be undergoing sinonasal surgery for this condition
* Diagnosis of CRS without NP and will be undergoing sinonasal surgery for this condition
* No diagnosis of CRS and NP and will be undergoing nasal surgery (septoplasty/rhinoplasty, nasal fracture repair,etc.)

Exclusion Criteria:

* Ages younger than 18 years and ages older than 70 years
* Diagnosis of an established immunodeficiency, pregnancy, coagulation disorder, a diagnosis of allergic fungal sinusitis (AFS), or cystic fibrosis
* Those with CRS with or without NP in whom systemic steroid therapy would be contraindicated
* Those who are dependent on systemic steroid therapy for sinonasal disease or any other condition

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Alterations of inflammatory cells, levels of key antibodies and cytokines, and expression of key epithelial genes | Prior to surgery and steroid treatment and day of surgery w/ or w/o having been treated w/ steroids

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Schleimer, PhD, Principal Investigator — Northwestern University and Northwestern Memorial Hospital
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Van Zele T, Claeys S, Gevaert P, Van Maele G, Holtappels G, Van Cauwenberge P, Bachert C. Differentiation of chronic sinus diseases by measurement of inflammatory mediators. Allergy. 2006 Nov;61(11):1280-9. doi: 10.1111/j.1398-9995.2006.01225.x. PMID 17002703
- [Background] Kanai N, Denburg J, Jordana M, Dolovich J. Nasal polyp inflammation. Effect of topical nasal steroid. Am J Respir Crit Care Med. 1994 Oct;150(4):1094-100. doi: 10.1164/ajrccm.150.4.7921442.
- [Background] Lavigne F, Cameron L, Renzi PM, Planet JF, Christodoulopoulos P, Lamkioued B, Hamid Q. Intrasinus administration of topical budesonide to allergic patients with chronic rhinosinusitis following surgery. Laryngoscope. 2002 May;112(5):858-64. doi: 10.1097/00005537-200205000-00015. PMID 12150618
- [Background] Wright ED, Agrawal S. Impact of perioperative systemic steroids on surgical outcomes in patients with chronic rhinosinusitis with polyposis: evaluation with the novel Perioperative Sinus Endoscopy (POSE) scoring system. Laryngoscope. 2007 Nov;117(11 Pt 2 Suppl 115):1-28. doi: 10.1097/MLG.0b013e31814842f8. PMID 18075447
- [Background] Meltzer EO, Hamilos DL, Hadley JA, Lanza DC, Marple BF, Nicklas RA, Adinoff AD, Bachert C, Borish L, Chinchilli VM, Danzig MR, Ferguson BJ, Fokkens WJ, Jenkins SG, Lund VJ, Mafee MF, Naclerio RM, Pawankar R, Ponikau JU, Schubert MS, Slavin RG, Stewart MG, Togias A, Wald ER, Winther B; Rhinosinusitis Initiative. Rhinosinusitis: developing guidance for clinical trials. J Allergy Clin Immunol. 2006 Nov;118(5 Suppl):S17-61. doi: 10.1016/j.jaci.2006.09.005. PMID 17084217
- [Background] Richer SL, Truong-Tran AQ, Conley DB, Carter R, Vermylen D, Grammer LC, Peters AT, Chandra RK, Harris KE, Kern RC, Schleimer RP. Epithelial genes in chronic rhinosinusitis with and without nasal polyps. Am J Rhinol. 2008 May-Jun;22(3):228-34. doi: 10.2500/ajr.2008.22.3162. PMID 18588753
- [Background] Kato A, Peters A, Suh L, Carter R, Harris KE, Chandra R, Conley D, Grammer LC, Kern R, Schleimer RP. Evidence of a role for B cell-activating factor of the TNF family in the pathogenesis of chronic rhinosinusitis with nasal polyps. J Allergy Clin Immunol. 2008 Jun;121(6):1385-92, 1392.e1-2. doi: 10.1016/j.jaci.2008.03.002. Epub 2008 Apr 14. PMID 18410958
- [Background] Xu G, Mou Z, Jiang H, Cheng L, Shi J, Xu R, Oh Y, Li H. A possible role of CD4+CD25+ T cells as well as transcription factor Foxp3 in the dysregulation of allergic rhinitis. Laryngoscope. 2007 May;117(5):876-80. doi: 10.1097/MLG.0b013e318033f99a. PMID 17473687
- [Background] Schleimer RP, Kato A, Kern R, Kuperman D, Avila PC. Epithelium: at the interface of innate and adaptive immune responses. J Allergy Clin Immunol. 2007 Dec;120(6):1279-84. doi: 10.1016/j.jaci.2007.08.046. Epub 2007 Oct 18. PMID 17949801
- [Background] Kato A, Schleimer RP. Beyond inflammation: airway epithelial cells are at the interface of innate and adaptive immunity. Curr Opin Immunol. 2007 Dec;19(6):711-20. doi: 10.1016/j.coi.2007.08.004. Epub 2007 Oct 24. PMID 17928212
- [Background] Kato A, Favoreto S Jr, Avila PC, Schleimer RP. TLR3- and Th2 cytokine-dependent production of thymic stromal lymphopoietin in human airway epithelial cells. J Immunol. 2007 Jul 15;179(2):1080-7. doi: 10.4049/jimmunol.179.2.1080. PMID 17617600
- [Background] Schleimer RP, Lane AP, Kim J. Innate and acquired immunity and epithelial cell function in chronic rhinosinusitis. Clin Allergy Immunol. 2007;20:51-78. PMID 17534045
- [Background] Kato A, Truong-Tran AQ, Scott AL, Matsumoto K, Schleimer RP. Airway epithelial cells produce B cell-activating factor of TNF family by an IFN-beta-dependent mechanism. J Immunol. 2006 Nov 15;177(10):7164-72. doi: 10.4049/jimmunol.177.10.7164. PMID 17082634
- [Background] Conley DB, Tripathi A, Seiberling KA, Schleimer RP, Suh LA, Harris K, Paniagua MC, Grammer LC, Kern RC. Superantigens and chronic rhinosinusitis: skewing of T-cell receptor V beta-distributions in polyp-derived CD4+ and CD8+ T cells. Am J Rhinol. 2006 Sep-Oct;20(5):534-9. doi: 10.2500/ajr.2006.20.2941. PMID 17063750
- [Background] Lane AP, Truong-Tran QA, Schleimer RP. Altered expression of genes associated with innate immunity and inflammation in recalcitrant rhinosinusitis with polyps. Am J Rhinol. 2006 Mar-Apr;20(2):138-44. PMID 16686375
- [Background] Anand VK, Kacker A, Orjuela AF, Huang C, Manarey C, Xiang J. Inflammatory pathway gene expression in chronic rhinosinusitis. Am J Rhinol. 2006 Jul-Aug;20(4):471-6. doi: 10.2500/ajr.2006.20.2891. PMID 16955782
- [Background] Schleimer RP. Glucocorticoids suppress inflammation but spare innate immune responses in airway epithelium. Proc Am Thorac Soc. 2004;1(3):222-30. doi: 10.1513/pats.200402-018MS. PMID 16113438
- [Background] Zhang N, Truong-Tran QA, Tancowny B, Harris KE, Schleimer RP. Glucocorticoids enhance or spare innate immunity: effects in airway epithelium are mediated by CCAAT/enhancer binding proteins. J Immunol. 2007 Jul 1;179(1):578-89. doi: 10.4049/jimmunol.179.1.578. PMID 17579079
- [Background] Bolger WE, Joshi AS, Spear S, Nelson M, Govindaraj K. Gene expression analysis in sinonasal polyposis before and after oral corticosteroids: a preliminary investigation. Otolaryngol Head Neck Surg. 2007 Jul;137(1):27-33. doi: 10.1016/j.otohns.2007.01.023. PMID 17599560
- See also: Principal Investigator Site — https://www.nm.org/doctors/search-results?terms=schleimer#all-1